CLINICAL TRIAL: NCT02108119
Title: The Effect of Probiotics on Symptoms and Intestinal Flora in Patients With Irritable Bowel Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Probi AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO008
Record Dates: First submitted 2014-04-01; First posted 2014-04-09 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Probiotics (Active Comparator)
  Interventions: Dietary Supplement: Probiotics
- Control placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Control placebo

INTERVENTIONS:
Dietary Supplement: Probiotics
  Arms: Probiotics
Dietary Supplement: Control placebo
  Arms: Control placebo

SUMMARY:
To demonstrate benefit of a probiotic product in adults with irritable bowel syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent
* Age ≥18 and ≤70 years at Visit 1
* IBS according to the Rome III criteria
* A score on abdominal pain NRS ≥3 and ≤6 at least two days a week measured the weeks before Visit 2 (baseline)
* IBS-SSS ≥75 and ≤300 at Visit 2 (baseline)
* Ability and willingness to understand and comply with the study procedures

Exclusion Criteria:

* Known intolerance or allergy to milk products (protein or lactose) or gluten
* History of alcohol or substance abuse six months prior to screening
* Known Hepatitis B or C or Human Immunodeficiency Virus (HIV) 1 or 2
* Female patients: currently pregnant or breast-feeding or intending to become pregnant during the study
* Abnormal results of the screening laboratory tests clinically relevant for study participation, as judged by the Investigator
* Other gastrointestinal disease(s) that explains the patient's symptoms, as judged by the Investigator
* Other severe disease(s) such as malignancy, severe coronary disease, kidney disease or neurological disease, as judged by the Investigator
* Symptoms indicating other severe disease(s) such as gastrointestinal bleeding, loss of weight or fever, as judged by the Investigator
* Severe psychiatric disease as judged by the Investigator
* Lack of suitability for participation in the study for any reason as judged by the Investigator
* Use of other probiotic products from Visit 1 and throughout the study.
* Consumption of antibiotic drugs 1 month prior to screening and throughout the study.
* Consumption of drugs on a regular basis which could interfere with symptom evaluation as judged by the Investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2014-05-02 (Actual); Primary Completion 2015-11-30 (Actual); Study Completion 2015-11-30 (Actual)

PRIMARY OUTCOMES:
Abdominal pain | 28 days
  0-10 numeric rating scale (NRS)

CONTACTS AND LOCATIONS:
Locations (1):
- PreCare Trial & Recruitment, Beek, Netherlands